CLINICAL TRIAL: NCT06499779
Title: Prescription of Valproate and Derivatives in Women of Childbearing Age: Qualitative Study
Acronym: VALPRO
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9135
Record Dates: First submitted 2024-07-05; First posted 2024-07-12 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Psychiatric Disorder
Keywords: Psychiatric disorder; Valproate
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The prescription of valproate in women of childbearing age has decreased by 82% in France, for mood disorders. Exposure to valproate during pregnancy 60%. However, the ANSM sent an alert document in August 2022 because there are still patients on valproate. In addition, there were 32 births taking valproate to mothers with bipolar disorder in 2018. The risks of exposure during pregnancy which occur in 10% of exposure cases are: congenital malformations; neurodevelopmental disorders including autism spectrum disorders, attention deficit disorders more or less hyperactivity, language disorders, motor disorders, mental delays; reduction in social, attentional, motor and language abilities; a lower level of education.

ELIGIBILITY:
Inclusion Criteria:

* Subject (≥16 years old)
* Female gender
* Prescription of Valproate and/or derivatives (Sodium Divalproate, Valpromide, Valproic Acid, Sodium Valproate) in an indication of psychiatric disorder for the period from January 1, 2021 to December 31, 2022,
* Subject not opposing, after information, the reuse of their data for the purposes of this research
* Holders of parental authority who do not object, after information, to the reuse of their child's data for the purposes of this research

Exclusion criteria:

* Subject and/or holder of parental authority having expressed opposition to participating in the study
* Impossibility of providing the subject with informed information (difficulties in understanding the subject, etc.)

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subject female (≥16 years old) having prescription of Valproate and/or derivatives (Sodium Divalproate, Valpromide, Valproic Acid, Sodium Valproate) in an indication of psychiatric disorder for the period from January 1, 2021 to December 31, 2022,
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-01-02 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05-02 (Estimated)

PRIMARY OUTCOMES:
Cause of valproate prescription in women of childbearing age | Up to 2 years
  Calculation of percentages, mean, median, standard deviation The results will be considered significant at the 5% threshold.

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Psychiatrie 2 - CHU de Strasbourg - France, Strasbourg, France